CLINICAL TRIAL: NCT03569215
Title: Psychiatric Disorders Among Egyptian Women With Prolonged Infertility With or Without Invitro Fertilization /Intracytoplasmic Spem Injection Failure
Brief Title: Psychiatric Disorders With Prolonged Infertility
Status: Completed | Type: Observational
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Ayman S Dawood, MD, Lecturer, Tanta University
Other Study IDs: Ayman
Record Dates: First submitted 2018-06-14; First posted 2018-06-26 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-08

CONDITIONS: Psychiatric Disorder; Invitro Fertilization /Intracytoplasmic Spem Injection Failure
MeSH Terms: conditions — Mental Disorders | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- IVF/ICSI failure: These patients had prolonged infertility with one or more failure of IVF/ICSI cycles
  Interventions: Behavioral: Questionnaire
- Prolonged infertility only: These patients had prolonged infertility without any trials of IVF/ICSI cycles
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — All included patients will be exposed to questionnaires and psychiatric diagnostic tests
  Other Names: Psychiatric diagnostic tests

SUMMARY:
Psychiatric disorders in women with prolonged infertility with or without IVF/ICSI failure will be included then a questionnaire will be applied plus psychiatric examinatins

DETAILED DESCRIPTION:
All patients will be recruited from both psychiatry and obstetrics and gynecology departments. Referred cases from gynecologists and Assisted reproductive technologies centers were also included.

Inclusion criteria:

Infertile couples Infertility >= 5 years invitro fertilization /intracytoplasmic spem injection failure for group 1 and not included for group 2

ELIGIBILITY:
Inclusion Criteria:

* Infertile women
* prolonged infertility ≥ 5 years
* Failed invitro fertilization /intracytoplasmic spem injection for group 1
* not bearing any children
* accepting to share in the study.

Exclusion Criteria:

* patients with diagnosed psychiatric or neurologic disorders
* patients with diabetes mellitus or any anatomical defects in genital tract
* patients who didn't complete their questionnaires.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — based on ID presentation
Study Population: All infertile women with prolonged infertility with or without history of IVF/ICSI failure
Sampling Method: Probability Sample
Enrollment: 324 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Prevalence and types of psychiatric disorders among prolonged infertility couples | 6 months
  Incidence and most common types of psychiatric disorders

CONTACTS AND LOCATIONS:
Overall Officials: Ayman Dawood, MD, Study Director — Lecturer at Tanta University; Reham Amer, MD, Principal Investigator — Lecturer at Tanta University
Locations (1):
- Reham Amer, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No
Individual participant data is secret as privacy and security of data is a must